CLINICAL TRIAL: NCT01648166
Title: A Population-based Case-control Study of Lung Cancer in Appalachian Kentucky: The Role of Environmental Carcinogens
Brief Title: Study of Lung Cancer in Appalachian Kentucky: The Role of Environmental Carcinogens
Status: Completed | Type: Observational
Sponsor: Susanne Arnold (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Susanne Arnold, MD, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: DOD2011-193
Record Dates: First submitted 2012-04-16; First posted 2012-07-24 (Estimated); Results first posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Lung Cancer
Keywords: trace; element; lung; cancer; Appalachia
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, live lymphocytes, serum, plasma, radon test kit, urine, water, soil, toenails, and hair.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- lung cancer cases: subjects with lung cancer who are greater than 17 years of age and live in Appalachian Kentucky
  Interventions: Other: Environmental sampling
- control subjects: subjects without lung cancer, greater than 17 who reside in Appalachian Kentucky
  Interventions: Other: Environmental sampling

INTERVENTIONS:
Other: Environmental sampling — Soil, water, blood, urine, hair and radon testing in homes in Appalachia

SUMMARY:
This is a research study about the relationship between lung cancer and environmental risk factors. The purpose of this study is to try to understand the effects of trace elements such as arsenic and chromium, as well as radon on the development of lung cancer. To do this, the investigators will collect information and environmental and biologic specimens from people who live in Appalachian Kentucky who a) have lung cancer or b) don't have lung cancer and will serve as control subjects. The investigators will create a specimen repository of from these people and their residences to compare differences in many risks factors for cancer. By doing this study, the investigators hope to learn why there are more lung cancers in Kentucky's fifth Congressional District than anywhere else in the nation.

DETAILED DESCRIPTION:
Appalachian Kentucky has one of the highest incidence rates of lung cancer in the United States. The disproportionately high incidence is not explained by tobacco alone. Preliminary analysis of trace element content in toenail samples reveals higher levels of arsenic, chromium and nickel in Appalachian Kentucky residents than elsewhere in Kentucky. Trace elements are known to promote carcinogenesis by increased oxidative stress, inflammation, DNA damage, and reduced DNA repair efficiency. These findings justify further investigation of the role that trace elements play in the development of lung cancer in this region. Hypothesis: The unexpectedly high rate of lung cancer in Appalachian Kentucky is associated with exposure to environmental carcinogens that increase oxidative stress and DNA damage.

Specific Aims Aim 1: Conduct a case-control study of lung cancer and matched controls in the 5th Congressional District of Kentucky to compare rates of moderate to high arsenic in lung cancer cases and controls.

Aim 2: Create a specimen repository of biologic and environmental samples from these subjects and their residences for analysis of DNA repair markers and, in the future, markers of oxidative stress and inflammation.

Aim 3: Fund four pilot projects which will utilize collected data from Aim 1 to develop investigators focused on lung cancer research in this study population and to generate preliminary data that will lead to independent funding.

Study Design: This is a population-based, case-control study encompassing the 5th Congressional District of Kentucky.

Relevance: This translational research and repository will fundamentally improve our understanding of the causes of the disproportionately high incidence of lung cancer in Appalachian Kentucky, foster collaboration among scientists dedicated to the study of lung cancer and provide a permanent resource to be used for future research.

ELIGIBILITY:
The following eligibility criteria are required for study entry and participation.

Inclusion (Lung cancer cases):

* Living persons with histologically or cytologically confirmed primary carcinoma of the lung (International Classification of Diseases-9, 162.2-162.9) between October 17, 2011 and October 16, 2013
* Age greater than 17
* Must be residents of the 5th Congressional District
* No prior history of any cancer (other than stage I and II non-melanomatous skin cancer)
* Must have a working phone
* Ability to participate in an in-person interview
* English speaking will be eligible for the study (no proxy respondents will be used)

Inclusion (Control cases):

* Age greater than 17
* No prior history of any cancer (other than stage I and II non-melanomatous skin cancer)
* Must be residents of the 5th Congressional District at the time they are matched to the case.
* Must have a working phone
* Ability to participate in an in-person interview
* English speaking will be eligible for the study (no proxy respondents will be used)

Exclusion:

* History of any cancers other than those listed above
* Non-residents of the 5th congressional district of Kentucky
* Age 17 years or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This case-control study will be performed in Appalachian Kentucky, specifically the 5th Congressional District of Kentucky and will include male and female subjects from the subset of all histologically or cytologically confirmed primary carcinoma of the lung (International Classification of Diseases-9, 162.2-162.9) over the age of 17 years old that occur in the 5th District between October 17, 20011 and November 14, 2013.
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne M Arnold, MD, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lung Cancer Cases | Control Subjects
Started | 153 | 367
Completed | 100 | 267
Not Completed | 53 | 100
Not completed — inadequate toenail samples | 53 | 100

BASELINE CHARACTERISTICS:
Population: population with trace element data available from toe nail analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Lung Cancer Cases | Control Subjects | Total
Number analyzed (Participants) | 100 | 267 | 367
Age, Continuous [Median (Full Range); unit: years] | 62 [39 to 89] | 62 [26 to 91] | 62 [26 to 91]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: only those with adequate toenails could complete the primary outcome measure of arsenic in nail.
  Participants
    Female | 61 | 148 | 209
    Male | 39 | 119 | 158
Region of Enrollment [Number; unit: participants]
  United States | 100 | 267 | 367

OUTCOME MEASURES:

1. Primary Outcome: Rate of Moderate to High Arsenic Level in Cases and Controls
Description: Conduct a case-control study of lung cancer and matched controls in the 5th Congressional District of Kentucky to compare rates of moderate to high arsenic in lung cancer cases and controls (primary endpoint).
Time Frame: up to three years
Population: those with adequate toenail arsenic concentrations
Measure: Median (Inter-Quartile Range); unit: mcg/dL
Arm/Group | Lung Cancer Cases | Control Subjects
Number analyzed (Participants) | 100 | 267
mcg/dL | 0.04 [0.03 to 0.06] | 0.04 [0.02 to 0.07]

ADVERSE EVENTS:
Arm/Group | Lung Cancer Cases | Control Subjects
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/267
Other Adverse Events (participants affected / at risk) | 0/100 | 0/267

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No